CLINICAL TRIAL: NCT02062424
Title: Diet and Prevention of Ischemic Heart Disease: a Translational Approach
Acronym: DIPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Denmark (Other)
Collaborators: University of Aarhus (Other); Harvard School of Public Health (HSPH) (Other); University of Copenhagen (Other); Ministry of Food, Agriculture and Fisheries, Denmark (Unknown)
Responsible Party: Principal Investigator, Inge Tetens, Professor, Technical University of Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Protocol no.:H-1-2013-110
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Ischemic Heart Disease
Keywords: ischemic heart disease, dietary guidelines
MeSH Terms: conditions — Myocardial Ischemia | interventions — 4',6-bis(2'imidazolinyl-4',5'-H)-2-phenylindole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DIPI: Danish national dietary guidelines (Active Comparator): The subjects will receive dietary advice according to the current national dietary guidelines
  Interventions: Other: DIPI
- DIPI: Specific IHD dietary guideline (Active Comparator): The subjects will receive dietary advice, according to the specific ischemic heart disease dietary guidelines.
  Interventions: Other: DIPI
- Normal dietary habits (No Intervention): The Subjects will be instructed to follow their normal dietary habits

INTERVENTIONS:
Other: DIPI
  Arms: DIPI: Danish national dietary guidelines; DIPI: Specific IHD dietary guideline

SUMMARY:
The objective of this study is to test the effect of substitution dietary guidelines that are specifically aimed at the prevention of ischemic heart disease (IHD) on the dietary intake in the general Danish population.

DETAILED DESCRIPTION:
225 participants will be included in the intervention. The intervention is planned to run for six months in a real life setting.

The study is a randomized, parallel dietary intervention study. Dietary intake, selected IHD biomarkers and anthropometric measurements will be measured at two visits during the intervention period as well as 6 months after the end of the intervention. The study includes a baseline visit followed by a visit where web based dietary records will be completed by the subjects and blood samples and anthropometrics will be measured.

The intervention will consist of information on dietary advice due to the specific IHD dietary guideline or the current national dietary guidelines. The information will be provided to the participants via leaflets and recipes.

After the baseline visit the subjects will be randomized to group A, B or C: In group A the subjects will receive dietary advice, according to the specific IHD dietary guideline, in group B the subjects will receive dietary advice according to the current national dietary guidelines and in group C the subjects will be instructed to follow their normal dietary habits.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women aged 30 to 65 years who has one or more self-assessed ischemic heart disease risk factors at screening: physical inactivity, overweight or obese (BMI ≥ 25/m2 ), waist circumference (≥ 80 cm for women, ≥ 94 cm for men). In addition, the participants should have the motivation and willingness to be randomized to any of the three groups, and to do their best to follow the given protocol .

Exclusion Criteria:

* no internet access or no access to a computer, smoking, pregnancy, or breast-feeding or planning to become pregnant within the next 12 months, a history of cardiovascular disease, type 2 diabetes, chronic disease / disorders that may affect the results of the study, substance abuse within the past 12 months, regular alcohol consumption > 21 units / week for men or > 14 units/ week for women, allergy or intolerance to food groups in the dietary guidelines, supplements with mega doses of nutrients that can have potential impact on ischemic heart disease risk markers (eg . fish oils).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Dietary intake | 6 month
  Dietary intake will be measured at two visits during the intervention period as well as 6 months after the end of the intervention.

SECONDARY OUTCOMES:
Selected ischemic heart disease biomarkers and anthropometric measurements | 6 month
  Selected IHD biomarkers and anthropometric measurements will be measured at two visits during the intervention period as well as 6 months after the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Tetens, Professor, Principal Investigator — Technical University of Denmark
Locations (1):
- Technical University of Denmark, Søborg, Denmark, Denmark

REFERENCES:
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 Aug 21;8(8):CD011737. doi: 10.1002/14651858.CD011737.pub3. PMID 32827219
- [Derived] Hooper L, Martin N, Jimoh OF, Kirk C, Foster E, Abdelhamid AS. Reduction in saturated fat intake for cardiovascular disease. Cochrane Database Syst Rev. 2020 May 19;5(5):CD011737. doi: 10.1002/14651858.CD011737.pub2. PMID 32428300
- [Derived] Arentoft JL, Hoppe C, Andersen EW, Overvad K, Tetens I. Associations between adherence to the Danish Food-Based Dietary Guidelines and cardiometabolic risk factors in a Danish adult population: the DIPI study. Br J Nutr. 2018 Mar;119(6):664-673. doi: 10.1017/S0007114517003695. Epub 2018 Jan 21. PMID 29352831